CLINICAL TRIAL: NCT01526681
Title: A Multicenter, Registry Study of Avance® Nerve Graft Utilization, Evaluations and Outcomes in Peripheral Nerve Injury Repair
Brief Title: Registry of Avance® Nerve Graft's Utilization and Recovery Outcomes Post Peripheral Nerve Reconstruction
Acronym: RANGER®
Status: Active, not recruiting | Type: Observational
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-CP-005
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Nerve Injuries
Keywords: Sensory Nerve; Mixed Nerve; Motor Nerve; Neurotization; Nerve Injury; Peripheral Nerve Injury
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Nerve Transfer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RANGER: Avance Nerve Graft: Processed Human Nerve Graft
  Interventions: Other: Processed Human Nerve Graft
- Historical Control for Standard Treatment: Literature review for outcomes from standard treatments, i.e. Autogenous Nerve Graft.
  Interventions: Other: Standard Treatment, Autogenous Nerve Graft, Direct Suture, etc.
- MATCH Arm: Contemporary Control: Addendum 1: Autogenous Nerve Graft and Nerve Tube Conduit
  Interventions: Other: Autogenous Nerve Graft; Device: Nerve Tube Conduit
- Sensation-NOW Arm: Breast Neurotization: Addendum 2: Post-mastectomy autologous breast reconstruction with or without neurotization
  Interventions: Procedure: Autologous Breast Reconstruction with Neurotization; Procedure: Autologous Breast Reconstruction without Neurotization

INTERVENTIONS:
Other: Processed Human Nerve Graft — Implantation of appropriate length of processed human nerve graft at the time of surgery
  Groups: RANGER: Avance Nerve Graft
Other: Standard Treatment, Autogenous Nerve Graft, Direct Suture, etc. — Historical control from established literature
  Groups: Historical Control for Standard Treatment
Other: Autogenous Nerve Graft — Nerve gap reconstructions with autogenous nerve graft within the upper extremity
  Groups: MATCH Arm: Contemporary Control
Device: Nerve Tube Conduit — Nerve gap reconstructions with nerve tube conduit within the upper extremity
  Groups: MATCH Arm: Contemporary Control
Procedure: Autologous Breast Reconstruction with Neurotization
  Groups: Sensation-NOW Arm: Breast Neurotization
Procedure: Autologous Breast Reconstruction without Neurotization
  Groups: Sensation-NOW Arm: Breast Neurotization

SUMMARY:
This study is a registry of general use of Avance Nerve Graft and is intended to evaluate the uses, response rates, and safety of Avance Nerve Graft in the real-life clinical setting. Optional addendums 1 and 2 included in the protocol are intended to establish comparative groups and focused subgroups within the registry.

DETAILED DESCRIPTION:
This is a multicenter registry study to collect utilization, safety, and outcomes data from medical record chart review of nerve reconstruction procedures throughout the body with Avance® Nerve Graft.

Addendum 1 (MATCH) establishes a comparative arm to collect data on nerve injuries repaired with nerve autografts and nerve tube conduits at select RANGER® participating sites.

Addendum 2 (Sensation-NOW) establishes a focused arm to collect data on autologous breast reconstructive procedures where neurotization was completed. Post-mastectomy autologous breast reconstruction procedures without neurotization will serve as an internal control group to allow for comparisons.

ELIGIBILITY:
Primary Study Criteria (RANGER Avance):

Inclusion Criteria:

* Males and Females who have undergone nerve repair using the Avance® Nerve Graft for the repair of a nerve injury
* Returned for at least one post-operative follow-up visit

Exclusion Criteria:

• Subject who in the opinion of the investigator, have not or likely will not complete at least some portion of the investigator's recommended follow-up.

Addendum 1 (MATCH) Criteria:

Inclusion Criteria:

* Have nerve transection injuries to the upper extremity;
* Have undergone tension free end to end nerve coaptation on both the proximal and distal portion of the nerve gap with nerve autograft or nerve entubulation with nerve tube conduit at a participating ANG-CP-005 registry site after 2004 and;
* Have completed sufficient follow-up assessments at a regeneration rate of 2mm/day to determine the outcomes of the repair or is willing to comply with site specific post-operative care procedures and assessments to determine the outcome of the repair.

Exclusion Criteria:

* Direct nerve repairs;
* Nerve gaps greater than 70mm;
* Subjects who, in the opinion of the investigator, were non-compliant to the investigator's post-operative treatment or rehabilitation instructions;
* Any subject who at the discretion of the Investigator is not suitable for inclusion in the study.

Addendum 2 (Sensation-NOW) Criteria:

Inclusion Criteria:

* Female ≥ 18 years old
* Undergo post mastectomy autologous breast reconstruction with one type of autologous flap (no stacked reconstructions or use of implant with autologous flap)
* Neurotization must be completed using a donor nerve from the flap and a recipient nerve from the chest
* Complete Sensory Assessment Testing with Semmes Weinstein Monofilaments (SWMF) and the following Breast-Q Questionnaires 60 - 120 days post-reconstruction:

  * Breast-Q Physical Well Being of the Chest
  * Breast-Q Satisfaction with Breast
  * Breast-Q Physical Well Being of the Abdomen
  * Breast-Q Abnormal Breast Sensations
  * Breast-Q Impact of Breast Sensation on Quality of Life
  * Breast-Q Return of Breast Sensation
* Able to provide informed consent and are willing to comply with post-operative care procedures and assessments

Exclusion Criteria:

* Surgical history of secondary revision surgery for partial or total flap loss
* Bilateral reconstruction with non-uniform treatment (i.e. 1 reconstructed breast is non-neurotized, 1 reconstructed breast is neurotized)
* Currently prescribed medication known to impact nerve regeneration or to cause peripheral neuropathy
* Currently undergoing IV chemotherapy or radiation
* Any subject who at the discretion of the Investigator is not suitable for inclusion in the study or is unlikely to comply with follow-up schedule

Additional Eligibility criteria to Modules

Module 1: Native Skin Reconstructions with and without neurotization.

* Buried flap reconstructions from nipple sparing mastectomy or skin sparing mastectomy OR a breast reconstruction from a skin sparing mastectomy with exposed flap skin in the peri-areolar region.
* Sensory assessments must be completed on ≥ 8 Zones of Native Skin.

  * Center zone measurement may be on either Native Skin or Flap Skin.
  * All Inner and Outer zone measurements must be on Native Skin.
  * De-identified photo of the breast reconstruction with 9 zones identified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects surgically repaired with Avance Nerve Graft to reconstruct peripheral nerve discontinuities.
Sampling Method: Non-Probability Sample
Enrollment: 3126 (Actual)
Dates: Start 2008-11; Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Avance Nerve Graft: Incidence of Avance Nerve Graft Related Adverse Events | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed through the course of their recovery based on Physician's standard of care practice or until lost to follow-up.
RANGER and MATCH: Sensory Function as measured by Medical Research Council Classification (MRCC) for sensory recovery | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for a change in sensory function, if applicable, of the reconstructed peripheral nerve through the course of their follow-up using Physician's standard of care sensory assessments or until lost to follow-up.
RANGER and MATCH: Motor Function as measured by Medical Research Council Classification (MRCC) for motor recovery | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for a change in motor function, if applicable, to the reconstructed peripheral nerve through the course of their follow-up using Physician's standard of care motor assessments or until lost to follow-up.
Sensation-NOW- Breast Neurotization: Sensory Function Post Autologous Breast Reconstruction | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for change in sensation through the course of their recovery using Physician's standard of care assessments or until lost to follow-up. Standard of care sensory assessment includes evaluation using Semmes Weinstein Monofilament kit measured in g/mm2.
Sensation-NOW- Breast Neurotization: Quality of Life Measurement Post Autologous Breast Reconstruction | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for change in quality of life as measured by Breast Q through the course of their recovery or until lost to follow-up using Physician's standard of care assessments. Standard of care assessments may include evaluation of quality of life via other scales or may be qualitatively documented.
Incidence of conduit, autograft, or procedure related adverse events | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed through the course of their recovery based on Physician's standard of care practice or until lost to follow-up.

SECONDARY OUTCOMES:
Pain Level | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for a change in pain level as measured by VAS, when available, through the course of their recovery using Physician's standard of care assessments for pain or until lost to follow-up.
RANGER and/or MATCH: Quality of Life Following Reconstruction of Peripheral Nerve | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for change in quality of life as measured by Disabilities of the Arm Shoulder and Hand Questionnaire (DASH), if available, through the course of their recovery or until lost to follow-up using Physician's standard of care assessments. Standard of care assessments may include evaluation of quality of life via other scales or may be qualitatively documented.
Cost of Care | Through study completion or until lost to follow-up, approximately 3 years
  Participants will be followed for cost of care, as converted to USD, from the surgical nerve procedure through the course of their recovery or until lost to follow-up using available data in the medical record from Physician's standard of care.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (46):
  - RANGER & MATCH: Arizona Center for Hand Surgery, Phoenix, Arizona
  - RANGER: Phoenix Children's Hospital, Phoenix, Arizona
  - RANGER & MATCH: University of California - Irvine, Orange, California
  - RANGER & MATCH: The Buncke Clinic, San Francisco, California
  - Sensation-NOW: Stanford University, Stanford, California
  - Sensation-NOW: University of Colorado School of Medicine, Aurora, Colorado
  - Sensation-NOW: George Washington University, Washington D.C., District of Columbia
  - RANGER: University of Miami, Miami, Florida
  - RANGER & MATCH: Florida Orthopaedic Institute, Tampa, Florida
  - RANGER: Hand & Upper Extremity Center of Georgia/Children's Hospital of Atlanta, Atlanta, Georgia
  - RANGER & MATCH: University of Kansas Medical Center, Kansas City, Kansas
  - Sensation-NOW: University of Kansas Medical Center, Kansas City, Kansas
  - RANGER: University of Kentucky, Lexington, Kentucky
  - Sensation-NOW: Advanced Reconstructive Care, LLC, Metairie, Louisiana
  - RANGER: Johns Hopkins University, Baltimore, Maryland
  - Sensation-NOW: Johns Hopkins University, Baltimore, Maryland
  - RANGER: Walter Reed National Military Medical Center, Bethesda, Maryland
  - MATCH: Hennepin County Medical Center, Minneapolis, Minnesota
  - RANGER & MATCH: University of Missouri - Columbia, Columbia, Missouri
  - Sensation-NOW: University of Nebraska Medical Center, Omaha, Nebraska
  - Sensation-NOW: University of Nevada, Las Vegas, Las Vegas, Nevada
  - RANGER: Multi-Disciplinary Specialists, Rutherford, New Jersey
  - RANGER & MATCH: OrthoCarolina Research Institute, Inc., Charlotte, North Carolina
  - RANGER: Duke University, Durham, North Carolina
  - RANGER: University of Cincinnati, Cincinnati, Ohio
  - Sensation-NOW: University of Cincinnati, Cincinnati, Ohio
  - RANGER: Cleveland Clinic, Cleveland, Ohio
  - RANGER: Ohio State University Medical Center, Columbus, Ohio
  - Sensation-NOW: Ohio State University Medical Center, Columbus, Ohio
  - Sensation-NOW: University of Pennsylvania, Philadelphia, Pennsylvania
  - Sensation-NOW: East Cooper Plastic Surgery, Mt. Pleasant, South Carolina
  - RANGER & MATCH: Campbell Clinic, Germantown, Tennessee
  - RANGER & MATCH: Vanderbilt University, Nashville, Tennessee
  - Sensation-NOW: Vanderbilt University, Nashville, Tennessee
  - Sensation-NOW: University of Texas Southwestern Medical Center, Dallas, Texas
  - RANGER: University of North Texas/John Peter Smith Hospital, Fort Worth, Texas
  - Sensation-NOW: University of North Texas/John Peter Smith Hospital, Fort Worth, Texas
  - Sensation-NOW: Baylor College of Medicine, Houston, Texas
  - Sensation-NOW: Houston-Methodist Central, Houston, Texas
  - Sensation-NOW: Houston-Methodist West/North, Houston, Texas
  - RANGER: Texas Tech University HSC, Lubbock, Texas
  - Sensation-NOW: Joshua Lemmon, MD, PLLC, Richardson, Texas
  - RANGER: San Antonio Military Medical Center, San Antonio, Texas
  - Sensation-NOW: PRMA Plastic Surgery, San Antonio, Texas
  - Sensation-NOW: Virginia Commonwealth University, Richmond, Virginia
  - RANGER & MATCH: University of Washington, Seattle, Washington
- RANGER: University Hospital, Vienna, Austria
- RANGER: North York General Hospital, Toronto, Ontario, Canada
- RANGER & MATCH: University Hospital Birmingham, England, Edgbaston, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No